CLINICAL TRIAL: NCT02549287
Title: Comparative Effectiveness Trail to Reduce Child Maltreatment, Improve Client Outcomes and Examine Client Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Whitaker (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Daniel Whitaker, Faculty Sponsor Investigator, Georgia State University
Organization: Georgia State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90CU0062
Record Dates: First submitted 2015-08-27; First posted 2015-09-15 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Child Maltreatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SafeCare (Experimental): SafeCare, an evidence-based home visiting program
  Interventions: Behavioral: SafeCare
- Supportive Case Management (Active Comparator): Child welfare services as usual
  Interventions: Behavioral: Supportive Case Management

INTERVENTIONS:
Behavioral: SafeCare — An evidence-based home visiting program
  Arms: SafeCare
Behavioral: Supportive Case Management — Child welfare services as usual
  Other Names: Services as Usual
  Arms: Supportive Case Management

SUMMARY:
In child welfare services, structured behavioral parenting programs have been documented to reduce important child-welfare outcomes, including child maltreatment recidivism.1-3 In this study, we attempt to learn which factors impacted implementation of an evidence-based practice (EBP) in a diversity of child-welfare serving sites and systems. The primary aim of this study was to identify and assess barriers and facilitators of implementation of a structured behavioral parenting program (SC). We utilized a qualitative research strategy that included semi-structured interviews and focus groups with several levels of staff responsible for implementing the model: program administrators, supervisors, and frontline staff (providers). Our second aim was to understand parent and provider reactions to SafeCare (SC) services and Supportive Case Management (SCM), especially parents' perceptions related to trajectory of burden, engagement, satisfaction, and perceived impact across intervention receipt. We employed mixed methods (both quantitative and qualitative data collection) to inform this question. Specifically, we (1) conducted qualitative interviews with families at two time points during the course of service, (2) collected session-by-session ratings from families on service reaction (perceived burden satisfaction, perceived effectiveness) and providers on family engagement, and (3) collected organizational environment surveys from providers at two time points. The final aim of this study wass to examine the short-term impact of SC versus SCM on client-centered outcomes. Quantitative surveys collected in the family's home at the beginning and end of services measured parenting variables, parent mental health and well-being, and child behavioral, social, and emotional well-being.

DETAILED DESCRIPTION:
The study design was a cluster randomized trial, with randomization occurring at the team level within each study site. We randomized providers within each site to be trained in SafeCare (n = 96) or to continue to deliver SCM (n = 96) which allowed us to control for site differences. From a statistical power perspective, it would have been preferable to randomize clients to interventions, but the fact that teams at community-based organizations typically served a defined geographic area would have meant that home visitors within each team would have had to deliver two distinct interventions raising the likelihood of cross-contamination which, in our experience, would have not been well managed by the study. Providers that were randomized were invited to participate in the study by completing a survey at baseline and 1-year follow-up which included measures of demographics, work experience, organizational factors (culture, climate, leadership) and individual attitudes and beliefs that may affect implementation and service quality. We recruited caregivers into the research study that were receiving services from randomized providers. Measurement of client-level outcomes were collected at baseline and 6-month follow up, as well as during service provision. Both quantitative and qualitative data were collected to capture both breadth and depth of family outcomes and experiences of the interventions.74 By focusing on measures of well-being, this study holds potential to expand the way in which the program effectiveness is conceptualized. This could be particularly important for dissemination of parenting programs to at-risk parents, who may be interested in different outcomes (e.g., improving their child's behavior) than child welfare systems, and findings may be useful for making interventions more appealing to consumers. To measure barriers and facilitators to implementing an evidence-based practice (EBP), we used a qualitative research strategy that included semi-structured interviews and focus groups with several levels of staff, responsible for implementing the model: program administrators, supervisors, and frontline staff (providers). This strategy would yield insight into an array of stakeholder perspectives concerning implementation. In contrast to most implementation studies, ours is the first to conduct a complementary set of interviews and focus groups with staff who have not been trained in SC, the SCM providers.

ELIGIBILITY:
Inclusion Criteria:

* Home Visitors: Home Visitors who are providing Supportive Case Management or being trained in SafeCare.
* Parents: English or Spanish speaking parents with a child between the ages of 0-5 years who are receiving services from a participating site.

Exclusion Criteria:

* Parents under the age of 18, who have no children under the age of 6 years, or do not speak English or Spanish will be excluded from this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Whitaker, PhD, Principal Investigator — Georgia State University
Locations (5):
- United States (5):
  - Southwest Iowa Family Access Center, Council Bluffs, Iowa
  - Children & Families of Iowa, Des Moines, Iowa
  - Mid Iowa Family Therapy Center, Des Moines, Iowa
  - Four Oaks, Iowa City, Iowa
  - Families First, Waterloo, Iowa

REFERENCES:
- [Derived] Whitaker DJ, Self-Brown S, Hayat MJ, Osborne MC, Weeks EA, Reidy DE, Lyons M. Effect of the SafeCare(c) intervention on parenting outcomes among parents in child welfare systems: A cluster randomized trial. Prev Med. 2020 Sep;138:106167. doi: 10.1016/j.ypmed.2020.106167. Epub 2020 Jun 20. PMID 32569643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were caregivers 18 or older, receiving services from a randomized provider, and had a child five or under. Participants were introduced to the study opportunity by their provider during a visit who referred interested participants to the Georgia State University-based research team to review the study procedures.
Units Other Than Participants: Team
Period: Overall Study
Arm/Group | SafeCare | Supportive Case Management
Started | 193; 17 Team | 96; 15 Team
Completed | 113; 17 Team | 64; 15 Team
Not Completed | 80; 0 Team | 32; 0 Team
Not completed — Lost to Follow-up | 65 | 26
Not completed — Withdrawal by Subject | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SafeCare | Supportive Case Management | Total
Number analyzed (Participants) | 193 | 96 | 289
Age, Categorical [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing Row population to differ from the Overall Population
  Participants
    number analyzed (Participants) | 191 | 94 | 285
    <=18 years | 2 | 1 | 3
    Between 18 and 65 years | 189 | 93 | 282
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data for 4 surveys were corrupted causing the Row population to differ from the Overall population
  years
    number analyzed (Participants) | 191 | 94 | 285
    (all) | 28.6 (6.9) | 31.5 (9.3) | 29.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing Row population to differ from the overall population
  Participants
    number analyzed (Participants) | 191 | 94 | 285
    Female | 159 | 88 | 247
    Male | 32 | 6 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing Row population to differ from the Overall population
  Participants
    number analyzed (Participants) | 191 | 94 | 285
    Hispanic or Latino | 11 | 8 | 19
    Not Hispanic or Latino | 178 | 84 | 262
    Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing Row population to differ from the Overall population
  Participants
    number analyzed (Participants) | 191 | 94 | 285
    American Indian or Alaska Native | 7 | 5 | 12
    Asian | 3 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 21 | 15 | 36
    White | 147 | 67 | 214
    More than one race | 1 | 2 | 3
    Unknown or Not Reported | 11 | 5 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Site 1 | 21 | 6 | 27
  United States: Site 2 | 2 | 5 | 7
  United States: Site 3 | 7 | 3 | 10
  United States: Site 4 | 42 | 5 | 47
  United States: Site 5 | 6 | 2 | 8
  United States: Site 6 | 19 | 2 | 21
  United States: Site 7 | 34 | 6 | 40
  United States: Site 8 | 23 | 27 | 50
  United States: Site 9 | 39 | 40 | 79
Education [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing Row population to differ from the Overall population. In addition, not all participants provided their level of education resulting in missing data.
  Participants
    number analyzed (Participants) | 191 | 93 | 284
    Less tha High School | 51 | 13 | 64
    High School | 64 | 36 | 100
    Some College | 76 | 44 | 120
Monthly Income [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing Row population to differ from the Overall population. In addition, not all participants provided information on their income resulting in missing data.
  Participants
    number analyzed (Participants) | 164 | 85 | 249
    < $600 | 62 | 24 | 86
    $600-$1250 | 55 | 29 | 84
    $1250 + | 47 | 32 | 79
Number of children in the home [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing Row population to differ from the Overall population. In addition, not all participants provided information on the number of children in their home resulting in missing data.
  Participants
    number analyzed (Participants) | 191 | 93 | 284
    No children in the home | 54 | 41 | 95
    1 child | 60 | 17 | 77
    2 children | 41 | 22 | 63
    3 or more childre | 36 | 13 | 49
Has a relationship partner [Count of Participants; unit: Participants] — Count of participants in a relationship with a partner. Population: Data for 4 surveys were corrupted causing the Row population to differ from the Overall population. In addition, not all participants provided information on relationship status.
  Participants
    number analyzed (Participants) | 188 | 92 | 280
    (all) | 119 | 43 | 162
Working [Count of Participants; unit: Participants] — Working full-time or part-time. Population: Data for 4 surveys were corrupted causing the Row population to differ from the Overall population.
  Participants
    number analyzed (Participants) | 191 | 94 | 285
    (all) | 89 | 51 | 140
Another caregiver in home [Count of Participants; unit: Participants] — Households that had another caregiver in the home. Population: Data for 4 surveys were corrupted causing the Row population to differ from the Overall population.
  Participants
    number analyzed (Participants) | 191 | 94 | 285
    (all) | 104 | 49 | 153
Alcohol use in the last 12 months [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing the Row population to differ from the Overall population. In addition, not all participants provided information on alcohol use history.
  Participants
    number analyzed (Participants) | 190 | 93 | 283
    (all) | 111 | 57 | 168
Illegal drug use in the last 12 months [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing the Row population to differ from the Overall population. In addition, not all participants provided information on illegal drug use history.
  Participants
    number analyzed (Participants) | 190 | 93 | 283
    (all) | 84 | 47 | 131
Victim of physical partner violence in the last 12 months [Count of Participants; unit: Participants] — Population: Data for 4 surveys were corrupted causing the Row population to differ from the Overall population. In addition, not all participants provided information on their physical partner violence history.
  Participants
    number analyzed (Participants) | 169 | 80 | 249
    (all) | 45 | 19 | 64

OUTCOME MEASURES:

1. Primary Outcome: Parenting Young Children Scale-Supporting Positive Behavior Sub-scale
Description: The Supporting Positive Behavior sub-scale of the Parenting Young Children Scale is made up of 7 items that assess supporting positive behavior (Example question: "Notice and praise your child's good behavior"). This subscale score is generated by calculating a mean of seven items on a 7-point scale (1=Not at all - 7=Almost Always). Theoretical range of means: 1-7; Actual range of means: 1-7. Higher scores represent higher degree of positive parenting skills. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring 6 or below were rated as low (n=125) and participants rating higher than 6 were rated as high (n=159).
Time Frame: Families were assessed at two time points: 1) after being invited into the study during a visit with their provider (Baseline) and, 2) approximately 6-months later (follow-up).
Population: Data for four surveys were corrupted causing the Row population to differ from the Overall population. In addition, Some participants missed or refused to answer questions.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 189 | 91
units on a scale
  Baseline | 6.14 [1 to 7] | 6.29 [3.14 to 7]
  6-month Follow-up: number analyzed (Participants) | 112 | 62
  6-month Follow-up | 6.43 [1.57 to 7] | 6.29 [1 to 7]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.12, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = 0.55, 95% CI 2-sided [-0.11 to 1.20]

2. Primary Outcome: Parenting Young Children Scale-Proactive Parenting Sub-scale
Description: The Proactive Parenting sub-scale of the Parenting Young Children Scale is made up of 7 items that assess proactive parenting (Example question: "Avoid struggles with your child by giving clear choices"). This subscale score is generated by calculating a mean of seven items on a 7-point scale (1=Not at all - 7=Almost Always). Theoretical range of means: 1-7; Actual range of means: 1-7. Higher scores represent higher degree of positive parenting skills. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring 6 or below were rated as low (n=148) and participants rating higher than 6 were rated as high (n=136).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 188 | 91
units on a scale
  Baseline: number analyzed (Participants) | 112 | 91
  Baseline | 5.79 [1 to 7] | 6.0 [1 to 7]
  6-month Follow-up: number analyzed (Participants) | 188 | 61
  6-month Follow-up | 6.29 [1 to 7] | 6.14 [1 to 7]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.14, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = 0.41, 95% CI 2-sided [-0.20 to 1.03]

3. Primary Outcome: Parenting Young Children Scale-Setting Limits Sub-scale
Description: The Setting limits sub-scale of the Parenting Young Children Scale is made up of 7 items that assess limit setting (Example question: "Stick to your rules and not change your mind"). This subscale score is generated by calculating a mean of seven items on a 7-point scale (1=Not at all - 7=Almost Always). Theoretical range of means: 1-7; Actual range of means: 1-7. Higher scores represent higher degree of positive parenting skills. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring 6.3 or below were rated as low (n=141) and participants rating higher than 6.3 were rated as high (n=143).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 188 | 91
units on a scale
  Baseline | 6.38 [1 to 7] | 6.57 [1 to 7]
  6-month Follow-up: number analyzed (Participants) | 112 | 61
  6-month Follow-up | 6.69 [1 to 7] | 6.57 [1 to 7]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.20, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = 0.44, 95% CI 2-sided [-0.20 to 1.07]

4. Primary Outcome: Parenting Stress Inventory - Short Form
Description: Parenting Stress Inventory - short form is a 36-item scale designed to measure stressors in parenthood including parental distress, dysfunctional interactions, and stressors related to having a difficult child. (Example question: "Sometimes I feel like my child doesn't like me and doesn't want to be close to me"). A total score generated by summing all 36 items on a 5-point scale (1=Strongly Agree - 5=Strongly Disagree). Theoretical total range: 36-180; Actual total range: 38-146. Lower scores represent more stress/dysfunction. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring 71 or below were rated as low (n=136) and participants rating higher than 71 were rated as high (n=148).
Time Frame: as for outcome 1
Population: Data for four surveys were corrupted causing the Row population to differ from the Overall population.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 191 | 93
units on a scale
  Baseline | 72 [40 to 152] | 74 [40 to 150]
  6-month Follow-up: number analyzed (Participants) | 113 | 62
  6-month Follow-up | 73 [41 to 140] | 74 [43 to 176]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.77, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = -0.07, 95% CI 2-sided [-0.58 to 0.43]

5. Primary Outcome: Protective Factors Survey-Parent Knowledge Sub-scale
Description: The Parent knowledge sub-scale of the Protective Factors is made up of 5 items that assess parent knowledge. (Example question: "There are many times when I don't know what to do as a parent"). This subscale score is generated by calculating a mean of 5 items on a 7-point scale (1=Never - 7=Always). Theoretical range of means: 1-7; Actual range of means: 3.4-7.0. Higher scores indicate higher parent knowledge. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring below 7 were rated as low (n=149) and participants rating 7 and higher were rated as high (n=133).
Time Frame: as for outcome 1
Population: Data for four surveys were corrupted causing the Row population to differ from the Overall population.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 191 | 91
units on a scale
  Baseline | 6.0 [3.4 to 7] | 6.0 [3.6 to 7]
  6-month Follow-up: number analyzed (Participants) | 111 | 62
  6-month Follow-up | 6.2 [3.4 to 7] | 5.9 [3.4 to 7]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.29, Marginal Model (e.g., GEE); Odds Ratio, log = 0.35, 95% CI 2-sided [-0.27 to 0.97]

6. Primary Outcome: Protective Factors Survey-Family Functioning Sub-scale
Description: The Family Functioning sub-scale of the Protective Factors is made up of 5 items that assess family functioning. (Example question: "My family pulls together when things are stressful"). This subscale score is generated by calculating a mean of 5 items on a 7-point scale (1=Never - 7=Always). Theoretical range of means: 1-7; Actual range of means: 1-7. Higher scores indicate higher family functioning. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring below 6 were rated as low (n=146) and participants rating 6 and higher were rated as high (n=133).
Time Frame: as for outcome 1
Population: Data for four surveys were corrupted causing the Row population to differ from the Overall population.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 188 | 91
units on a scale
  Baseline | 5.0 [1 to 7] | 5.0 [1 to 7]
  6-month Follow-up: number analyzed (Participants) | 110 | 62
  6-month Follow-up | 5.4 [1 to 7] | 5.2 [1 to 7]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.15, Marginal Model (e.g., GEE) — Other [Marginal Model (e.g., GEE)]; Odds Ratio, log = 0.49, 95% CI 2-sided [-0.08 to 1.06]

7. Primary Outcome: Brief Symptom Inventory-Significant Case Percentage
Description: The Brief Symptom Inventory is a 53-item scale designed to measure a range of emotional health states including depression, anxiety, somatization, and others. (Example question: "How much were you distressed by nervousness or shakiness inside"). The 'significant case' definition from the BSI was used and includes those with elevated scores (higher than 2) on any of the subscales. The percentage of participants that were considered a 'significant case' is reports. The 'case' definition from the BSI, which includes elevation on any of the subscale. The Brief Symptom Inventory is a 53-item scale designed to measure a range of emotional health states including depression, anxiety, somatization, and others. A total score or the, Global Severity Index, is generated by calculating a mean of all 53 items; lower scores indicate lower levels of distress.
Time Frame: as for outcome 1
Population: Data for four surveys were corrupted causing the Row population to differ from the Overall population.
Measure: Count of Participants; unit: Participants
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 191 | 93
Participants
  Baseline | 80 | 40
  6-month Follow-up: number analyzed (Participants) | 108 | 58
  6-month Follow-up | 36 | 23
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.61, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = -0.11, 95% CI 2-sided [-0.73 to 0.52]

8. Primary Outcome: BSI-Global Severity Index
Description: The Brief Symptom Inventory is a 53-item scale designed to measure a range of emotional health states including depression, anxiety, somatization, and others. (Example question: "How much were you distressed by nervousness or shakiness inside"). The Global Severity Index calculated a mean of all of the BSI subscales which includes 53 items on a 5-point scale (0=Not at all-4=Extremely). Theoretical range of means: 0-4; Actual range of means: 0.0-3.5). Higher scores indicate higher existence of symptoms. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, females scoring below .77 and males scoring below .57 were rated as low (n=197) and females rating .78 and higher and males rating .58 and higher were rated as high (n=87).
Time Frame: as for outcome 1
Population: Data for four surveys were corrupted causing the Row population to differ from the Overall population.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 191 | 93
units on a scale
  Baseline | 0.35 [0 to 3.54] | 0.42 [0 to 3.21]
  6-month Follow-up: number analyzed (Participants) | 112 | 62
  6-month Follow-up | 0.25 [0 to 3.38] | 0.37 [0 to 3.17]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.47, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = -0.22, 95% CI 2-sided [-0.76 to 0.32]

9. Primary Outcome: Devereaux Early Child Assessment-Initiative Sub-scale
Description: The Initiative sub-scale of the Devereaux Early Child Assessment (DECA) is made up of 11-18 items (depending on child's age) that assesses the child's initiative behavior. (Example question: "Did the child do things for himself"). This subscale score generates a t-score of standardized norms from a sum of the 11-18 items on a 5-point scale (0=Never - 4=Very frequently). Theoretical range of means: 28-72; Actual range of means: 28-72. Higher ratings represent a higher degree of child initiation. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring below 56 were rated as low (n=110) and participants rating 56 and higher were rated as high (n=118).
Time Frame: as for outcome 1
Population: Data for four surveys were corrupted causing the Row population to differ from the Overall population. In addition, Some participants missed or refused to answer questions. Lastly, errors in survey branching based on child's age required discarding those responses which reduced the total number of participants analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 157 | 71
units on a scale
  Baseline | 54.92 (11.62) | 54.97 (11.80)
  6-month Follow-up: number analyzed (Participants) | 78 | 44
  6-month Follow-up | 55.44 (11.20) | 55.84 (10.34)
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.65, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Slope = -0.75, 95% CI 2-sided [-3.70 to 2.20]

10. Secondary Outcome: Mother-Child Neglect Scale (MCNS)
Description: The Mother-Child Neglect Scale (MCNS) is a 22-item scale designed to assess caregiving behaviors in four domains: physical, cognitive, supervision, and emotional needs. (Example question: "I make sure my child sees a doctor when he/she needs one"). A total score generated by calculating a mean of the 22 items rated on a 4-point scale (1=Strongly Agree - 4=Strongly Disagree). Theoretical range of means: 1-4; Actual range of means: 1.2-3.9. Lower scores indicate less neglectful behaviors. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring 3.65 and below were rated as low (n=139) and participants rating higher than 3.65 were rated as high (n=145).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 190 | 93
units on a scale
  Baseline | 3.68 [1.2 to 3.95] | 3.64 [2.64 to 3.86]
  6-month Follow-up: number analyzed (Participants) | 112 | 61
  6-month Follow-up | 3.71 [2.73 to 3.95] | 3.67 [2.64 to 3.95]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.64, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = 0.05, 95% CI 2-sided [-0.59 to 0.69]

11. Secondary Outcome: Confusion, Hubbub, and Order Scale (CHAOS)
Description: The CHAOS scale (Confusion, Hubbub, and Order) is a 15-item scale used to measure structure and chaos in the home environment. (Example question: "There is very little commotion in our home"). A total score generated by calculating a mean of all 15 items on a 4-point scale (1=Very much like your own home - 4=Not at all like your own home). Theoretical range of means: 1-4; Actual range of means: 1.0-2.7. Lower scores indicate less chaos. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring 1.5 or below were rated as low (n=151) and participants rating higher than 1.5 were rated as high (n=133).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 188 | 91
units on a scale
  Baseline | 1.47 [1 to 2.73] | 1.47 [1 to 2.50]
  6-month Follow-up: number analyzed (Participants) | 111 | 59
  6-month Follow-up | 1.53 [1 to 2.40] | 1.47 [1 to 2.60]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.44, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = -0.25, 95% CI 2-sided [-0.79 to 0.29]

12. Secondary Outcome: Family Resources Scale - Revised
Description: The Family Resources Scale - Revised is a 40-item scale that assesses the adequacy of family needs in four domains: basic needs, money, time for self, and time for family. (Example question: "How well is the following need being met: House or apartment"). A total count of resources needed out of 40 assessed. Resources were considered needed if the participant indicated the resource was 'Not at all' met, 'A little' met, or 'Sometimes' met (5-point scale: 1=Not at all - 5=Almost always). Theoretical range of means: 0-40; Actual range of means: 0-40. Higher ratings indicating a higher number of resources needed. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants with 9 or fewer needs not met were rated as low (n=152) and participants with 10 and higher needs not met were rated as high (n=132).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 190 | 92
units on a scale
  Baseline | 9.0 [0 to 37] | 9.0 [0 to 40]
  6-month Follow-up: number analyzed (Participants) | 112 | 62
  6-month Follow-up | 8.0 [0 to 39] | 6.5 [0 to 40]
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.47, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Odds Ratio, log = 0.25, 95% CI 2-sided [-0.39 to 0.89]

13. Primary Outcome: Devereaux Early Child Assessment-Attachment Sub-scale
Description: The Attachment sub-scale of the Devereaux Early Child Assessment (DECA) is made up of 8-18 items (depending on child's age) that assesses the child's attachment behavior. (Example question: "Did the toddler accept comfort from a familiar adult"). This subscale score generates a t-score of standardized norms from a sum of the 8-18 items on a 5-point scale (0=Never - 4=Very frequently). Theoretical range of means: 28-72; Actual range of means: 28-72. Higher ratings represent a higher degree of child attachment. Because the data were heavily skewed toward the positive end of the scale, the measure was dichotomized into high vs. low based on an approximate median split. Specifically, participants scoring below 52 were rated as low (n=101) and participants rating 52 and higher were rated as high (n=138).
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SafeCare | Supportive Case Management
Number analyzed (Participants) | 166 | 73
units on a scale
  Baseline | 52.4 (12.0) | 53.4 (12.16)
  6-month Follow-up: number analyzed (Participants) | 90 | 46
  6-month Follow-up | 53.8 (12.0) | 56.3 (11.3)
Statistical Analysis 1: Comparison: SafeCare vs Supportive Case Management; Intent-to-treat (ITT) framework (multiple imputation used), Multilevel model applied; Test type: Superiority; p = 0.63, Marginal Model (e.g., GEE) — Group by time interaction effect reported here; Slope = -0.18, 95% CI 2-sided [-3.57 to 3.22]

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-Cause Mortality was not monitored/assessed.
Arm/Group | SafeCare | Supportive Case Management
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/193 | 0/96
Other Adverse Events (participants affected / at risk) | 0/193 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT02549287/Prot_SAP_000.pdf